CLINICAL TRIAL: NCT06979492
Title: Prophylactic Transfusion In Pregnant in Women With Sickle Cell Disease
Acronym: ProTIP
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ross Fasano, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00007288
Record Dates: First submitted 2025-05-13; First posted 2025-05-20 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Sickle Cell Disease; Pregnancy Related
Keywords: Blood transfusion; Anemia
MeSH Terms: conditions — Anemia, Sickle Cell; Anemia | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Other): Patients randomized to the control group will receive standard care for SCD alone. As part of the standard of care, women with SCD who become pregnant and who are on hydroxyurea (HU) will have the HU suspended by their primary SCD provider.
  Interventions: Other: Control group
- Red Blood Cell (RBC) Transfusion (Experimental): Participants will receive a blood transfusion between 6 and 20 weeks of gestation. It will be repeated at 3-6 week intervals, aiming to maintain HbS <30%
  Interventions: Biological: Prophylactic Transfusion Intervention group: Transfusion

INTERVENTIONS:
Biological: Prophylactic Transfusion Intervention group: Transfusion — For participants randomized to the prophylactic transfusion intervention group, the first RBC transfusion will occur within 3 weeks of randomization. All transfusions will be managed per SOC.
  SOC prophylactic RBC transfusion management is as follows: transfusions are performed at 3-6 week intervals with the intent to maintain a pre-transfusion hemoglobin S level at <30%. All participants will have a complete blood count, reticulocyte count, hemoglobin fractionation, complete metabolic profile with LDH, ferritin, and type/screen at baseline and within 3 days of all monthly transfusions. All RBC transfusions must be compatible between the recipient and the donor and antigen matched for Rh (D/Cc/Ee) and Kell antigens at a minimum. For participants with a previous history of RBC alloimmunization, extended matched RBCs will be provided (Rh, Kell, Duffy, Kidd, S/s) per NHLBI/ASH guidelines to minimize further alloimmunization.
  Arms: Red Blood Cell (RBC) Transfusion
Other: Control group — Participants randomized to the control group will be followed per SOC. SOC management for pregnant women with SCD includes but is not limited to
  * Clinic appointments with an SCD provider every 2 months
  * Lab draws - complete blood count, reticulocyte count, hemoglobin fractionation, complete metabolic profile with LDH and ferritin.
  Arms: Standard of Care

SUMMARY:
The goal of this study is to determine if there is a positive effect of prophylactic red blood cell (RBC) transfusion of leukoreduced, ABO, Rh (D/Cc/Ee) and Kell matched blood compared to standard of care on the number of episodes of acute sickle cell disease (SCD) manifestations or pregnancy-related complications requiring acute health care encounters (acute care/ER/Hospital visits) or resulting in death over the entirety of pregnancy until 2 months post-partum in women with SCD.

RBC transfusion is the only disease-modifying therapy for pregnant women with SCD, and it is considered a standard treatment option however, there exists no consensus on the role of transfusion therapy in preventing SCD-related pregnancy complications.

Participants will be randomly assigned to repeated red blood cell transfusions or the standard of care. Participants will be on study for about 8-10 months (Pregnancy through 2 months post-partum).

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is a common genetic disorder that results from the homozygous presence of abnormal β-globin chains (hemoglobin Hb SS, Hb SC, HbSβ thalassemia). SCD causes red blood cells to become rigid, leading to various acute and chronic manifestations: chronic hemolytic anemia, poor growth, acute vaso-occlusive pain crises (VOC), priapism (in men) acute ischemic stroke, acute chest syndrome (ACS), and chronic organ damage within the spleen, kidneys, liver, lungs and heart.

High rates of both maternal and fetal morbidity and mortality complicate pregnancy in patients affected by SCD. SCD pregnancies have been linked to higher rates of obstetrical complications, including preeclampsia, venous thromboembolism, intrauterine growth restriction, preterm delivery, and small-for-gestational-age infants. In addition, sickle-related maternal complications are common during pregnancy. More than 50% of women with SCD have a VOC in the antenatal period (76% for HbSS vs 27% for Hb SC). ACS in pregnancy is seen in 7% to 20% of women with HbSS and approximately 5% in women with HbSC. Prophylactic transfusion therapy has established benefits in stroke prevention and preoperative optimization in SCD patients, but its use in pregnancy has not been established. Because hydroxyurea (HU) may be teratogenic, RBC transfusion is the only disease-modifying therapy available for pregnant women with SCD.

The decision to put a pregnant woman with SCD on chronic transfusion therapy is entirely based on provider preference and patient willingness. RBC transfusions are considered a standard treatment option for pregnant women with SCD and transfusion therapy widely used, however there exists no consensus among providers on the role of chronic transfusion therapy in preventing SCD-related pregnancy complications and no prospective randomized controlled study investigating the role of prophylactic transfusion for prevention of both maternal and fetal morbidity has been done.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Diagnosis of SCD of any genotype (i.e., HbSS, HbSC, HbSβ thalassemia)
* 18 Years and older
* Currently pregnant at 6 weeks through 20 weeks of gestation.
* Ability to understand the purposes and risks of the study and willingly give informed consent.
* For participants with private health insurance, insurance pre-approval for blood transfusions

Exclusion Criteria:

* Currently on chronic transfusion therapy before pregnancy
* Prior history of DHTR with hyperhemolysis
* Red cell antibody history, which would prevent the provision of adequate red cell units to support chronic transfusions.
* Unable or unwilling to receive blood transfusion for social, religious, or clinical reasons
* Known current triplet pregnancy
* Current diagnosis of major medical or psychiatric comorbidity, which in the randomizing clinician's opinion renders them unable to enter a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — This study aims to determine the optimal management of pregnant women with SCD. Researchers will only include the following special population: Pregnant women.
Enrollment: 50 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Hospital admissions rate | Baseline (enrollment) up to 8 weeks post-partum
  Number of participants who require hospital admission during study participation divided by the total number of participants. Collected from medical records
Number of maternal emergency department (ED)/Acute care visits | Baseline (enrollment) up to 8 weeks post-partum
  Collected from medical records
Number of SCD-related complications per group | Baseline (enrollment) up to 8 weeks post-partum
  Sickle cell complications (vaso-occlusive crisis (VOC) / acute chest syndrome (ACS) / cerebral stroke) collected from medical records
Number of participants with pregnancy related complications | Baseline (enrollment) up to 8 weeks post-partum
  Number of participants who will develop pregnancy-related complications (pre-eclampsia, venous thromboembolism, infection). Collected from medical records
Maternal death | From randomization up to 8 weeks post-partum
  Number of women who die at any gestational age during pregnancy or within 8 weeks after delivery from any cause arising from the pregnancy or its management, but not from incidental or accidental causes, divided by the total number of participants.

SECONDARY OUTCOMES:
Adult Sickle Cell Quality of Life Measurement System (ASCQ-Me) | 2, 4, 6, 8 and 10 months post randomization.
  The Adult Sickle Cell Quality of Life Measurement System (ASCQ-Me) is a validated patient-reported outcome measure of physical, mental, and social health in adults with SCD. Patient-reported outcome measure of pain level in the past 7 days. The ASCQ-Me pain scale ranges from 0-100, with a standardized sickle cell disease population mean of 50 (standard deviation=10), where lower scores signify worse disease impact. A modified version of the validated ASCQ-Me will be used.
Patient reported outcomes measurement information system (PROMIS) | 2, 4, 6, 8 and 10 months post randomization.
  The patient-reported outcomes will be assessed using a health-related quality of life questionnaire, a modified version of the validated sickle-cell specific quality of life instruments, PROMIS
  The PROMIS Short-Form scale is a generic measure of health-related quality of life (HRQL) that assesses physical, mental, and social health. It has a recall period of 7 days and yields separate Physical Health and Mental Health subscale scores, which range from 0 to 100 and are standardized to a US population mean of 50 and standard deviation (SD) of 10. Each question usually has five response options ranging in value from one to five. To find the total raw score for a short form with all questions answered, sum up the values of the responses to each question. For example, for the adult 8-item form, the lowest possible raw score is 8; the highest possible raw score is 40. For each subscale, a higher score connotes better functioning.
Infant birth weight | At delivery up to 42 weeks of pregnancy
  Infant's birth weight from medical records.
Preterm delivery | Up to delivery (36 weeks of pregnancy)
  Number of women delivered before 37 weeks gestational age divided by the total number of participants randomized.
APGAR Scores | 1 and 5 minutes after neonate's delivery
  The Apgar score is a scoring system doctors and nurses use to assess newborns after delivery. At most, a child will receive an overall score of 10. A score of 7 to 10 five minutes after birth is reassuring, 4 to 7 is moderately abnormal, and 0 to 3 is concerning. The Apgar scoring system is divided into five categories. Each category receives a score of 0 to 2 points.
  A: Activity/muscle tone P: Pulse/heart rate G: Grimace (response to stimulation, such as suctioning the baby's nose) A: Appearance (color) R: Respiration/breathing
Number of neonatal intensive care unit/critical care admissions | After neonate's delivery up to 1 week post-partum
  The neonate's admission to the intensive care unit/critical care admission will be documented from medical records.
Perinatal death | From 28 weeks of pregnancy up to 1 week post-partum
  Number of babies who died from 28 weeks gestational age up to seven days post-delivery (comprising all still births and early neonatal deaths divided by total births.
Fetal demise/stillbirth | From enrollment up to 42 weeks of pregnancy
  Fetal demise refers to the spontaneous intrauterine death of a fetus at any time during pregnancy.
Number of participants with new RBC alloantibodies | From enrollment up to 8 weeks post-partum
  Participants who have been assigned to receive chronic simple blood transfusions will have monthly labs prior to their scheduled transfusion as per SOC to assess for new alloantibodies.
Number of participants with transfusion reactions | From enrollment up to 8 weeks post-partum
  Participants will be carefully monitored for transfusion-related adverse events throughout the intervention phase of the study.
Number of participants with an increase in iron overload (serum ferritin) | From enrollment up to 8 weeks post-partum
  Transfusion iron burden will be monitored with monthly serum ferritin levels during the study, which is standard of care monitoring for patients undergoing chronic transfusion therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Fasano, MD, Principal Investigator — Emory University
Locations (1):
- Grady Health System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No